CLINICAL TRIAL: NCT01170559
Title: Use of Implantable Loop Recorders as a Primary Investigation of Infrequent Undiagnosed ArrhythmIa Symptoms in the Emergency Department
Brief Title: Use of Loop Recorders for Diagnosis of Palpitations in A&E
Acronym: LIAISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 006628 BLT
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2014-08

CONDITIONS: Palpitations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: ILR Group (Experimental): Group allocated to receiving an ILR in the A&E department.
  Interventions: Device: Implantable Loop Recorder
- Group 2: Conventional (No Intervention): Group randomised to conventional lines of investigation

INTERVENTIONS:
Device: Implantable Loop Recorder
  Other Names: Reveal XT
  Arms: Group 1: ILR Group

SUMMARY:
Heart rhythm abnormalities underlie one of the common presenting complaints to the A&E and out-patient departments, specifically awareness of heart beats or palpitations. Unless an ECG (electrocardiogram) tracing of the heart rhythm can be recorded while the patient is having symptoms, it is very difficult to determine the cause of the palpitations. The conventional approach is to refer these patients from the emergency departments to the Cardiology outpatients where they undergo repeated short term rhythm monitoring hoping to record the rhythm underlying the patient's complaint. Unfortunately, this often yields no results thus delaying definitive treatment and incurring extra costs of repeated investigations and A&E presentations. This study aims to compare the ability of the conventional approach to establish a definite diagnosis compared to that of an early invasive monitoring approach with a small implantable device that records the heart rhythm at all time for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Good history of episodic symptomatic sustained palpitations (sudden onset and offset, fast heart beats, may be associated with shortness of breath or dizziness)
* Terminates before presentation to hospital
* Episodes occur at a frequency of less than once every two weeks
* Never previously caught on ECG or ambulatory monitoring
* Normal resting ECG

Exclusion Criteria:

* Contraindication to ILR implantation i.e. ongoing oral anticoagulation with INR >1.6, ongoing infection, sepsis or fever, etc.
* Palpitations suggestive of extrasystoles (single missed or dropped beats)
* Known or suspected severe valvular or myocardial heart disease

  * An audible heart murmur
  * Any abnormality on the surface ECG
* Thyrotoxicosis
* Patients who refuse an ILR when offered will not be included in either limb of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2010-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the proportion of patients achieving a definite diagnosis in each of the two groups at the end of one year | 1 year

SECONDARY OUTCOMES:
The time taken from randomisation in the A&E to making the diagnosis (if any) in each group | 1 Year
The cost of achieving a diagnosis in each group | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, MD, FRCP, Principal Investigator — Barts and the London NHS Trust, Queen Mary University of London
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom